CLINICAL TRIAL: NCT03675165
Title: Can You Reduce Diabetes Symptomatology by Becoming Your 'Best Possible Self': The Role of Stress and Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Ben Gibson, Principal Investigator, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18/NSP/067
Record Dates: First submitted 2018-09-04; First posted 2018-09-18 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Prevention; Psychology; Self-Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive a tailored version of Laura King's 'Best Possible Self' intervention: a brief, self-administered, psychological intervention. It is fundamentally a writing exercise, whereby recipients are asked to spend 10 minutes writing about their best possible future self and the steps they need to take to become that person. This helps the individual set goals while facilitating positive affect. Our version of the task has people focus on their health-related goals in particular.
  Interventions: Behavioral: Best Possible Self
- Waiting List Control (No Intervention): Participants are informed that they are on a waiting list and will receive the intervention at the end of the study.

INTERVENTIONS:
Behavioral: Best Possible Self — A writing exercise developed in 2001 by Laura King. The frequency of engagement with the exercise is down to the user's discretion though we recommend to them to write things down once every week for the duration of the study.
  Other Names: Best Possible Selves
  Arms: Intervention

SUMMARY:
The purpose of this study is to examine how the 'Best Possible Self' (BPS) intervention influences diabetes symptomatology over a four week period by assessing stress and resilience as mediatory effects. Half of the participants will receive the BPS straight away while the other half will be put on a waiting list and will act as the control group.

DETAILED DESCRIPTION:
The BPS is a "positive" psychology intervention; i.e. it facilitates positive emotion in order to achieve psychological, behavioural, and even physiological changes. The present team's previous research has demonstrated that the BPS is effective at reducing certain diabetes symptoms, though the exact mechanisms by which it does so are unclear. According to the Stress Buffering Model of Physical Activity, psychological stress is the catalyst that triggers behavioural and physiological responses critical to health while positive emotions can improve health by helping people to cope. The Broaden and Build Theory of Positive Emotions, meanwhile, suggests that this is because positive emotions allow people to build resilience.

In this study, the aim is to examine whether stress and resilience in particular mediate the relationship between intervention and diabetes symptoms. Research around stress and resilience has shown these factors to be important not only in the physical health of people with diabetes but for also decreasing illness symptomatology in non-clinical samples more generally.

ELIGIBILITY:
Inclusion Criteria:

* Non-clinical sample
* 18+
* Access to the internet

Exclusion Criteria:

* Severe mental illness (such as schizophrenia or bipolar depression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Diabetes Symptomatology (assessed using the Diabetes Symptoms Checklist - Revised) | Four Weeks
  Subscales assess the existence of, and the distress caused by, fatigue, cognitive, pain, sensory, cardiology, ophthalmology, hypoglycaemia, and hyperglycaemia symptoms individually. For each sub-scale, participants can score between 0 and 5, with a lower score meaning fewer symptoms and less distress caused by that subset of symptoms. Subscales do not come together to create a total symptomatology score.

OTHER OUTCOMES:
Self-Reported Stress (assessed using the Perceived Stress Scale) | Four weeks
  Mediatory Effect. Individual scores are added up and can range from 0-40. A higher score means that the individuals perceives themselves to be more stressed.
Self-Reported Resilience (assessed using the Six-Item Brief Resilience Scale) | Four Weeks
  Mediatory Effect. Responses are added up to give a score between 6 and 30. The total sum is then divided by 6 (the number of questions). A higher score indicates a higher level of resilience.
Diabetes Risk (calculated using the Canadian Diabetes Risk Questionnaire) | Four Weeks
  Control Variable. A total risk score is assessed by summing up the scores of each of the 12 questions. Scores range from 0-87. A lower score indicates less risk. Participants with a score of < 21 are low risk, participants with a score of 21 - 32 are medium risk, and participants with a score of >32 are high risk.

CONTACTS AND LOCATIONS:
Overall Officials: Kanayo F Umeh, Study Director — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual participant data.

REFERENCES:
- See also: Study link — https://ljmupsych.qualtrics.com/jfe/form/SV_41SfG1puMuBJHEN

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03675165/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03675165/ICF_001.pdf